CLINICAL TRIAL: NCT05998785
Title: A Multi-Center, Prospective Case Series Evaluating Insertional Achilles Tendinopathy Repair Augmented with TAPESTRY® Biointegrative Implant
Brief Title: Embody Insertional Achilles Tendinopathy
Acronym: IAT
Status: Terminated | Type: Observational
Why Stopped: Administrative issues with IRB, none of which impacted the health/safety/welfare of the subjects, has resulted in enrollment suspension and subsequent study termination.
Sponsor: Zimmer Biomet (Industry)
Collaborators: Embody Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EMBODY-002
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Insertional Achilles Tendinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: TAPESTRY Biointegrative Implant — Collagen-based implant composed of type I bovine collagen and poly(D,L-lactide). It is designed to function as a non-constricting, protective layer between the tendon and surrounding tissues. Preclinical studies of the Tapestry implant showed dense collagenous fibrous connective tissue ingrowth into and around the implant.

SUMMARY:
The primary objective of this study is to evaluate the long-term effects on ankle/Achilles tendon pain after repair of insertional Achilles tendinopathy (IAT) augmented with TAPESTRY Biointegrative Implant.

DETAILED DESCRIPTION:
This study is a prospective case series of patients who have had insertional Achilles tendinopathy repair augmented with the Tapestry Biointegrative Implant. The primary aim of the study is to describe patient reported pain 12 months after surgical repair with Tapestry. The secondary aims are to assess the proportion of study subjects that experience treatment-related adverse events post-surgery, treatment related serious adverse events resulting in second surgical intervention, quality of life and other patient reported outcomes at all follow up timepoints post-surgery, and tissue thickness measured with MRI at 6 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 21 years and older;
* Insertional Achilles tendonitis requiring surgery that has failed at least 2 weeks of conservative management, which consist of:

  1. Shoe modification; or
  2. Nonsteroidal anti-inflammatory drugs; or
  3. Physical Therapy with/without modalities.
* Chronic Achilles tendon pain lasting longer than 3 months;
* MRI of the ankle within 30 days prior to the study surgery;
* Ability and willingness to comply with prescribed post-operative rehabilitation program;
* Ability and willingness to comply with follow-up regimen;
* Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures; and
* Ability to read, understand, and complete subject-reported outcomes in English.

Exclusion Criteria:

* History of Achilles tendon rupture;
* Previous Achilles tendon surgery on the index ankle;
* Genetic collagen disease, hypersensitivity, or objection to using bovine-derived materials;
* History of auto-immune or immunodeficiency disorders;
* History of chronic inflammatory disorders;
* Oral steroid use in last 2 months or injectable steroid use in last 4 weeks;
* History of heavy smoking (> 1 pack per day) within last 6 months;
* Hypersensitivity to poly(D,L-lactide) materials;
* Metal implants, fillings, shrapnel, and/or screws;
* Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study;
* Currently involved in any injury litigation or worker's compensation claims relating to the index ankle;
* Enrolled, or plans to enroll, in another clinical trial during this studythat would affect the outcomes of this study; or
* History of non-compliance with medical treatment, physical therapy/rehabilitation, or clinical study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrolled subjects will include adults with insertional Achilles tendonitis requiring surgery, who meet the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Pain/VAS | 12 months post-surgery
  Visual Analog Scale (VAS) survey

SECONDARY OUTCOMES:
Safety/Adverse Events | Surgery, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks, 3 months, 6 moths and 12 months post-op
  * Procedure and/or treatment related adverse events;
  * Procedure and/or treatment related Serious Adverse Events (SAE)
  * Procedure and/or treatment related Serious Adverse Events (SAE) necessitating a second surgical intervention (SSI);
Patient Satisfaction | 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks, 3 months, 6 moths and 12 months post-op
  Patient Satisfaction Survey
Return to Normal Activity | 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks, 3 months, 6 moths and 12 months post-op
  Return to Normal Activity survey
AOFAS | Baseline, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks, 3 months, 6 moths and 12 months post-op
  American Orthopedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot questionnaire
SF-12 | Baseline, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks, 3 months, 6 moths and 12 months post-op
  12-item Short Form- Health Survey
Tissue Thickness | Baseline and 6 months post-op
  MRI tissue thickness of the Achilles tendon at baseline and 6 months post-surgery. Tissue thickness will be measured by trained personnel per the EMBODY-002 MRI procedure manual.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weil Foot and Ankle Institute, Libertyville, Illinois
  - Utica Park Clinic, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No